CLINICAL TRIAL: NCT05859490
Title: A Phase I/II Study Of The Immunogenicity Of The Yellow Fever Vaccine 17D (YFVax®) In Adults With Prior 17D Vaccination
Brief Title: Immunogenicity of Yellow Fever Vaccine 17D in Adults With Prior 17D Vaccination
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, William Messer, Associate Professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00025307
Record Dates: First submitted 2023-04-05; First posted 2023-05-16 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Yellow Fever; Immunization; Infection
Keywords: 17D; vaccination; immunity
MeSH Terms: conditions — Yellow Fever; Infections

STUDY DESIGN:
Intervention Model Description: All subjects receive the same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Vaccination arm (Experimental): Participants will receive a standard dose of of the yellow fever vaccine 17D (YFVax(r)), 0.5mL suspension in normal saline administered subcutaneously once.
  Interventions: Biological: 17D

INTERVENTIONS:
Biological: 17D — Vaccine administration in subjects previously vaccinated with 17D.
  Other Names: YFVax

SUMMARY:
The goal of this clinical trial is to assess the immune response to the yellow fever vaccine 17D in adults with prior 17D vaccination. The main questions this study aims to answer are:

* how does prior vaccination affect antibody responses to re-vaccination?
* how does prior vaccination affect the immune cell response to re-vaccination?

Participants will:

* have been previously vaccinated with 17D.
* be re-vaccinated with 17D.
* provide medical and travel histories.
* provide a blood sample prior to vaccination
* provide a blood sample approximately every other day for 14 days after vaccination.
* provide a blood sample approximately 28 days after vaccination.
* complete a daily diary of symptoms following vaccination for 14 days.
* report any additional symptoms after 14 days.

DETAILED DESCRIPTION:
In this study the investigators use 17D revaccination as a live-virus challenge to test the hypothesis that neutralizing antibody titers correlate with YFV protection. The investigators will prospectively characterize pre-boost antibodies titers, vaccine viremia, acute immune responses and post-boost titers in vaccinees receiving boost 17D vaccinations. The investigators expect to identify neutralizing antibody titers above which sterilizing immunity is conferred and titers below which it is not. These Aims will set a foundation for future studies to further dissect determinants of 17D and other live-attenuated vaccine induced immunity and establish metrics that could allow efficient prioritization of 17D vaccination and optimize 17D use in the face of current and future outbreaks.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥20 to <50 years.
2. Male or female.
3. In good health at the time of screening as determined by medical history, physical examination, and clinical judgement of the investigator.
4. Documented history of Yellow fever vaccination 8 or more years prior. Documentation must be on a primary (not copied) vaccination card or a fully completed electronic medical record entry including date of administration and lot number administered.
5. Subjects who can comply with all trial procedures and are available for the duration of follow-up.

Exclusion Criteria:

1. A clinically active infection or self-reported body temperature ≥38°C (100.4°F) within 3 days of scheduled date of vaccination (consider whether the finding is an exclusion criterion or criterion for delay of vaccination see Section 8.3).
2. A known hypersensitivity or allergy to any of the trial vaccine components including eggs.
3. Behavioral/cognitive impairment that, in the investigator's opinion, may interfere with the subject's ability to participate safely in the trial.
4. Any history of neurologic disorder, seizure disorder or neuro-inflammatory disease.
5. Any illness, or history of any illness that, in the investigator's opinion, could interfere with the trial or pose an additional risk to the subject during the trial period.
6. Known or suspected impairment/alteration of immune function, including:

   1. Chronic use of oral steroids within 60 days prior to enrollment. Inhaled steroids are allowed.
   2. Receipt of parenteral steroids within 60 days prior to screening visit.
   3. Receipt of immunoglobulins and/or any blood products within the 3 months prior to enrollment or planned receipt during the trial.
   4. Receipt of immunostimulants within 60 days prior to screening visit
   5. Immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within 6 months of enrollment.
   6. Known Human Immunodeficiency Virus (HIV) infection or HIV-related disease.
   7. Hepatitis C virus infection.
   8. Genetic immunodeficiency.
7. History of splenic or thymic dysfunction.
8. Any serious chronic or progressive disease as assessed by the investigator (eg, neoplasm, hematologic malignancies, insulin dependent diabetes; cardiac, renal, or hepatic disease).
9. Body Mass Index (BMI) greater than or equal to 35 kg/m2.
10. Concurrent participation in any clinical trial with another investigational product 30 days prior to or during the conduct of this trial.
11. Vaccination within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrollment or plans to receive any vaccine within 28 days of trial vaccine administration (consider whether applicable as an exclusion criterion or criterion for delay of trial vaccine administration).
12. Use of antipyretics and/or analgesic medications within 24 hours prior to vaccination. Trial entry should be delayed to allow for a full 24-hours to have passed since last use of antipyretics and/or analgesic medications (consider whether applicable as an exclusion criterion or criterion for delay of trial vaccine administration).
13. Subjects with history of substance or alcohol abuse within the past 2 years.
14. Subjects who are pregnant or breastfeeding.
15. Subjects of childbearing potential who are sexually active with men and have not used "acceptable contraceptive methods" for at least 2 months prior to enrollment.

    1. Of "childbearing potential" is defined as beyond onset of menarche and not: menopausal for 2 or more years, post bilateral tubal ligation at 1 year prior, post bilateral oophorectomy for at least 1 year or post hysterectomy.
    2. "Acceptable birth control methods" include:

    <!-- -->

    1. Hormonal contraceptives (such as oral, injection, transdermal patch, implant, cervical ring).
    2. Barrier method (condom with spermicide or diaphragm with spermicide) every time during intercourse.
    3. Intrauterine device.
    4. Monogamous relationship with vasectomized partner (partner must have been vasectomized for at least 6 months prior to the subject's enrollment.
16. Subjects of childbearing potential who are sexually active with men and refuse acceptable contraceptive method up to 28 days after the vaccination.
17. Any positive or indeterminate pregnancy test.
18. Planned vaccination (during the trial conduct) against any other vaccine preventable disease.
19. Planned travel (during the trial) to any YFV endemic area.
20. Screening serology consistent with prior history of dengue, zika, West Nile or Japanese encephalitis virus infection.

It may occur that a prospective subject meets all entry criteria except one that relates to short term clinical condition (e.g., fever, recent use of excluded medications). Under these circumstances, eligibility for delayed trial enrollment may be considered after inclusion/exclusion criteria have been rechecked, and if the subject is confirmed to be eligible.

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Neutralizing antibody titer boost following vaccination | 28 days
  four-fold rise in neutralization antibody titer before and after vaccinatioin
vaccine viremia following vaccination | 14 days
  detection of vaccine virus in subject blood

SECONDARY OUTCOMES:
CD4+ immune cell response to vaccination | 28 days
  Frequency of CD4+ cell populations on day 0, 2, 8, 14, and 28 post vaccination

OTHER OUTCOMES:
CD8+ immune cell response to vaccination | 28 days
  Frequency of CD8+ cell populations on day 0, 2, 8, 14, and 28 post vaccination
cytokine response to vaccination | 28 days
  Cytokine levels measured on days 0, 1, 2, 8, 14, and 28 days post vaccination
vaccine virus titer | 1 day
  quantity of vaccine virus in vaccine vial on vaccination day 0
Memory B cell response to vaccination | 28 days
  YFV specific memory B cell frequency on days 1, 2, 8, 14 and 28 days post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: William Messer, MD PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Coded samples and/or data will be made available to other researchers.
Supporting Information: Study Protocol
Time Frame: For up to 5 years after the completion of the study.
Access Criteria: The PI will review all sample and data requests. A request will include a scope of work and justification for the work. All approved requests will be conducted under an M/DTA.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT05859490/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-24): https://cdn.clinicaltrials.gov/large-docs/90/NCT05859490/ICF_001.pdf